CLINICAL TRIAL: NCT00559455
Title: Phase II Study of Oxaliplatin + 5-FluoroUracil/Leucovorin (Eloxatin+5-FU/LV) in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Phase II Study of Eloxatin+5-FU/LV in Patients With Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, Sanofi-aventis Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXALI_L_02859
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: Oxaliplatin — 85mg/m², 2 hours IV infusion, Day 1; Every 2 weeks
Drug: Fluorouracil — 400mg/m², 2 hours IV bolus, Day 1; 22 hours continuous IV infusion 600mg/m², Day 1 and Day 2; Every 2 weeks
Drug: Leucovorin — 200mg/m², Day 1 and Day 2; Every 2 weeks

SUMMARY:
Primary objective:

To determine the Tumor Response Rate of patients with hepatocellular carcinoma treated with the combination chemotherapy of Eloxatin+5-FU/LV

Secondary objective:

To evaluate time to progression, 6month survival, overall survival, safety and tolerability of patients with hepatocellular carcinoma treated with the combination chemotherapy of Eloxatin+5-FU/LV

ELIGIBILITY:
Lists of Inclusion and Exclusion criteria:

* Patients must have histologically confirmed hepatocellular carcinoma
* Patients must have measurable disease by CT scan
* Have not received previous palliative systemic chemotherapy for metastatic disease. (Adjuvant chemotherapy or radiation therapy for non target lesion can be allowed.)
* Patients progress after previous local treatment and at the time of randomization is at least 4 weeks after the last interventional therapy (Hepatic Artery Infusion, Trans-Artery Embolization or Trans-Artery Chemo-Embolization) or at least 4 weeks after the last radiotherapy/ablation/ Percutaneous Ethanol Injection to the target lesion.
* WHO 0-2 grades (Karnofsky Performance Score ≥ 70)
* Patients must have adequate organ and marrow function:

  * Neutrophilus ≥ 1.5 x 10^9/L
  * Platelets ≥ 75 x 10^9/L
  * Asparagine AminoTransferase, Alanine AminoTransferase < 2.5 x Upper Normal Limit(UNL)
  * Total Bilirubin ≤ 1.5 x UNL
  * International Normalized Ratio < 1.5
  * Child stage A or B
  * Creatinine ≤ 1.5 X UNL

Exclusion Criteria:

* Documented allergy to platinum compound or to other study drugs.
* Active Gastro-Intestinal bleeding and active haematologic malignancy
* Previous liver transplantation.
* Patients concomitantly receiving any other anti-cancer therapy.
* Patients who are receiving any other study treatments.
* Pregnant or lactating women or women of childbearing potential without proper contraceptive methods.
* History of other malignant diseases, except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix.
* Central nervous system metastasis
* Other serious illness or medical conditions
* Neuropathy ≥ grade 2

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Tumor Response Rate evaluated using RECIST (Response Evaluation Criteria in Solid Tumors) by physical examination, chest X-ray, abdomen-pelvis CT (Computed tomography) scan | every 6 weeks

SECONDARY OUTCOMES:
Time to Progression (TTP), 6 month survival, overall survival, AFP | from the signature of Informed Consent up to end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Hyang Rim Kim, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Seoul, South Korea